CLINICAL TRIAL: NCT05422196
Title: Evaluation of Computer-Guided Secondary Alveolar Cleft Bone Grafting With and Without Platelet-Rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A08080920
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Alveolar Bone Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No platelet-rich fibrin was added to the cleft site during grafting.
- Study group (Experimental): Platelet-rich fibrin was added to the cleft site during grafting.
  Interventions: Procedure: Platelet-rich fibrin

INTERVENTIONS:
Procedure: Platelet-rich fibrin — Addition of platelet-rich fibrin into the cleft site.
  Arms: Study group

SUMMARY:
This study aims at investigating the role of platelet-rich fibrin in alveolar cleft secondary grafting. This grafting is done from the patient's chin using a computer-guided stent that is customized for each patient, and the cleft volume is analysed at first to estimate the needed amount of bone to be harvested.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients who are classified according to the American Society of Anesthesiologists (ASA) physical status classification as class I.
2. Patients seeking treatment and accepting to be enrolled in the study, so as their guardians.
3. Patients who will age 9-14 years old by the surgery day.
4. Patients with adequate chin bone volume that could be harvested without marked donor site morbidity, as pre-determined by cone beam computed tomography.

Exclusion Criteria:

1. Patients with systemic illness, i.e. ASA(22) classes II, III, IV, and V.
2. Patients with previously operated alveolar clefts and seeking revision for the same cleft.
3. Patients that wouldn't be able to attend the recalls.
4. Patients with other craniofacial anomalies and associated syndrome conditions.
5. Edentulous maxilla, atypical or non-described cleft diagnosis.
6. Patients with history of chemotherapy or radiotherapy.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Closure of oronasal fistula | Ten days postoperatively
  * By questioning the patient if there's a nasal regurgitation or not.
  * Qualitative outcome (positive or negative).
Closure of oronasal fistula | Six months postoperatively
  * By questioning the patient if there's a nasal regurgitation or not.
  * Qualitative outcome (positive or negative).
Volume of newly formed bone | Six months postoperatively
  * By computerized measurement on the Cone-Beam Computed Tomography software. (Volume tool in Invesalius ® software (Invesalius, CTI, Brazil)).
  * Quantitative outcome (in cubic millimetres (mm3)).
Average density of newly formed bone | Six months postoperatively
  * By computerized measurement on the Cone-Beam Computed Tomography software. (Average density tool in Invesalius ® software (Invesalius, CTI, Brazil)).
  * Quantitative outcome (in Hounsfield Units (HU)).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Addakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided